CLINICAL TRIAL: NCT05152264
Title: High Frequency, High Intensity Transcutaneous Electrical Nerve Stimulation for Endometriosis-related Chronic Pain - a Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation for Endometriosis-related Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 274998
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis-related Pain
Keywords: Endometriosis; Chronic pain; Transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Endometriosis; Chronic Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Patients with frequent pain and high pain intensity (≥ 4 according to Numeric Rating Scale, NRS) will be randomized to additional treatment with TENS or conventional analgesic treatment for 8 weeks in order to evaluate the acute effects of TENS treatment (n=40). Patients with endometriosis-related pain that is not frequent or without high pain intensity constitute an external control group. All patients in the study will receive TENS treatment for a total of 16 weeks, for evaluation of long-term effects of TENS treatment in chronic endometriosis-related pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TENS (transcutaneous electrical nerve stimulation) (Active Comparator): Patients with endometriosis-related chronic frequent pain and high pain intensity (≥ 4 according to Numeric Rating Scale, NRS) randomized to transcutaneous electrical nerve stimulation as add-on treatment in addition to conventional analgesic treatment. Treatment with transcutaneous electrical nerve stimulation (TENS) during 16 weeks.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Conventional analgesic treatment (Active Comparator): Patients with endometriosis related chronic frequent pain and high pain intensity (≥ 4 according to Numeric Rating Scale, NRS) randomized to conventional analgesic treatment for 8 weeks. After 8 weeks the patients are treated with transcutaneous electrical nerve stimulation (TENS) during 16 weeks.
  Interventions: Other: Conventional analgesic treatment
- External control group (Active Comparator): Patients with endometriosis-related pain that is not frequent or without high pain intensity (< 4 according to Numeric Rating Scale, NRS) constitute an external control group. The patients are treated with transcutaneous electrical nerve stimulation as add-on treatment in addition to conventional analgesic treatment. Treatment with transcutaneous electrical nerve stimulation (TENS) during 16 weeks.
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Treatment with transcutaneous electrical nerve stimulation (TENS) during 16 weeks.
  Arms: External control group; TENS (transcutaneous electrical nerve stimulation)
Other: Conventional analgesic treatment — Conventional analgesic treatment. Conventional analgesic treatment may include no pharmacological treatment if the patient does not use any analgesics.
  Arms: Conventional analgesic treatment

SUMMARY:
The study evaluates the effect of TENS (transcutaneous electrical nerve stimulation) as add-on treatment compared with conventional analgesic treatment in patients with endometriosis-related chronic pain. Patients with frequent pain and high pain intensity will be randomized to additional treatment with TENS or conventional treatment for 8 weeks to evaluate the acute effects of TENS treatment (n=40). Patients with endometriosis-related pain that is not frequent or without high pain intensity constitute an external control group. All patients in the study will receive TENS treatment for a total of 16 weeks, for evaluation of long-term effects of TENS treatment.

DETAILED DESCRIPTION:
Endometriosis affects approximately one in ten women of childbearing age and may involve both acute pain related to the menstrual cycle and chronic pain. Usual analgesic therapy is often inadequate and/or involves unacceptable side effects and risks with long-term use. Transcutaneous electrical nerve stimulation (TENS) is a patient controlled treatment for pain relief with few side-effects. To date there is limited knowledge of how TENS treatment should be carried out for optimal pain relief in this patient group. The aim of the study is asses the effect of TENS as add-on treatment compared with conventional analgesic treatment in patients with endometriosis-related chronic pain. Patients with frequent pain and high pain intensity (≥ 4 according to Numeric Rating Scale, NRS) will be randomized to additional treatment with TENS or conventional treatment for 8 weeks in order to evaluate the acute effects of TENS treatment (n=40). Patients with endometriosis-related pain that is not frequent or without high pain intensity constitute an external control group. All patients in the study will receive TENS treatment for a total of 16 weeks, for evaluation of long-term effects of TENS treatment in chronic endometriosis-related pain. Prior to start of TENS treatment, all patients receive education on chronic endometriosis-related pain and TENS treatment. Study participants will be asked to participate in a qualitative follow-up within the study including a semi-structured individual interview (n=10-15) before intervention and a semi-structured focus group (n=9-15) interview after completion of TENS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Consents to participation in the study
* Verified endometriosis (by laparoscopy or ultrasound).
* Chronic endometriosis-related pain (> 3 months), available for TENS treatment
* Functioning, stable endometriosis-specific hormonal drug therapy. The endometriosis-specific drug therapy must be unchanged for the last 3 months and no gynecological surgical procedures for the treatment of endometriosis are planned during the next 7 months (during study participation). The endometriosis-specific drug therapy does not refer to analgesic therapy for symptom relief of endometriosis-related pain.

Exclusion Criteria:

* Patient with inability to understand and use written and spoken Swedish
* Patient with pacemaker and/or ICD or other electronic implants
* Patient with impaired sensation over the painful area
* Malignant disease with an expected survival <12 months
* Alcohol or substance abuse
* Serious untreated psychiatric illness and/or psychological condition that is the primary determinant of the patient's condition
* Participating in another intervention study with possible impact on current study outcome measures
* Patient who is using >90 morphine equivalents/day
* Patient who is electro-acupuncture
* Pregnancy

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 8 weeks after randomization
  Pain intensity according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to endometriosis-related chronic pain

SECONDARY OUTCOMES:
Pain intensity | 16 weeks after start of TENS treatment
  Pain intensity according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to endometriosis-related chronic pain
Physical activity | 16 weeks after start of TENS treatment
  Minutes of physical activity per week at moderate and vigorous intensity physical activity (MVPA), minutes of sedentary behaviour (SED) assessed by accelerometry
Self-assessed physical activity | 16 weeks after start of TENS treatment
  Minutes of physical activity per week (physical exercise and daily exercise) and minutes of sedentary behaviour per week.
Consumption of analgetics | 8 weeks after randomization
  Consumption of primary and secondary analgetics including opioid consumption in morphine equivalent doses
Consumption of analgetics | 16 weeks after start of TENS treatment
  Consumption of primary and secondary analgetics including opioid consumption in morphine equivalent doses
Change in pain intensity | 8 weeks after randomization
  Pain intensity according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to endometriosis-related chronic pain, Likert scale (1= "worse," 2= "unchanged," 3= "slightly improved," 4= "much improved," 5 = "very much improved,"and 6= "completely improved").
Change in pain intensity | 16 weeks after start of TENS treatment
  Pain intensity according to numeric rating scale (score from 0 to 10, where 0 is described as "no pain" and 10 as "worst pain imaginable") with regard to endometriosis-related chronic pain, Likert scale (1= "worse," 2= "unchanged," 3= "slightly improved," 4= "much improved," 5 = "very much improved,"and 6= "completely improved").
Health Related Quality of Life (HRQL) according to SF36 | 8 weeks after randomization
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) according to SF36 | 16 weeks after start of TENS treatment
  Assessed with RAND Short Form 36 (SF36). The 36 items in the questionnaire are grouped into eight subscale scores: physical functioning, role limitations caused by physical problems, bodily pain, general health, energy/vitality, social functioning, role limitations caused by emotional problems and mental health. The subscale scores range from 0-100, the higher score, the better health related quality of life.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 8 weeks after randomization
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Health Related Quality of Life (HRQL) assessed with EQ-5D | 16 weeks after start of TENS treatment
  Assessed with EQ-5D-5L. The questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Health Related Quality of Life (HRQL) assessed with EHP 30 | 8 weeks after randomization
  Assessed with Endometriosis Health Profile 30. The EHP score indicate the extent of self-reported ill health on each of the 5 domains measured (Pain, Control and powerlessness, Social support, Emotional well-being, Self-image). Each scale is standardised on a scale of 0 - 100, where 0 indicates the best health status through to 100 worst health status.
Health Related Quality of Life (HRQL) assessed with EHP 30 | 16 weeks after start of TENS treatment
  Assessed with Endometriosis Health Profile 30. The EHP score indicate the extent of self-reported ill health on each of the 5 domains measured (Pain, Control and powerlessness, Social support, Emotional well-being, Self-image). Each scale is standardised on a scale of 0 - 100, where 0 indicates the best health status through to 100 worst health status.
General Self-Efficacy Scale | 8 weeks after randomization
  The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life, Likert scale (1= Not at all true 2= Hardly true 3= Moderately true 4= Exactly true)
General Self-Efficacy Scale | 16 weeks after start of TENS treatment
  The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life, Likert scale (1= Not at all true 2= Hardly true 3= Moderately true 4= Exactly true)
Insomnia Severity | 8 weeks after randomization
  Total score from the 7-item Insomnia Severity Index where total score ranges from 0-28 and higher scores indicate greater severity of insomnia.
Insomnia Severity | 16 weeks after start of TENS treatment
  Total score from the 7-item Insomnia Severity Index where total score ranges from 0-28 and higher scores indicate greater severity of insomnia.
Days of sick-leave | 8 weeks after randomization
  Number of days of sick-leave
Days of sick-leave | 16 weeks after start of TENS treatment
  Number of days of sick-leave

OTHER OUTCOMES:
Anxiety, depression | 8 weeks after randomization
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Anxiety, depression | 16 weeks after start of TENS treatment
  Assessed with the Hospital Anxiety and Depression (HAD) scale. The scale consists of 14 items on a four-point response scale ranging from 0-3. Seven items for depression and 7 items for anxiety with a score range from 0-21. For each factor (anxiety or depression), the results are interpreted as follows: < 8 points indicates within normal range, 8-10 points indicates possible and >10 points indicates probable anxiety or depression.
Patient treatment satisfaction according to NRS | 8 weeks after randomization
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Patient treatment satisfaction according to NRS | 16 weeks after start of TENS treatment
  Self-reported treatment satisfaction with regard to pain relief, how acceptable the patient finds the treatment and hospital care. Numeric rating scale (score from 0 to 10, where 0 is described as "not satisfied at all" and 10 as "very satisfied") and numeric rating scale (score from 0 to 10, where 0 is described as "not acceptable at all" and 10 as "very acceptable").
Multidimensional Assessment of Interoceptive Awareness | 8 weeks after randomization
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is an 8-scale state-trait questionnaire with 32 items to measure multiple dimensions of interoception by self-report.
Multidimensional Assessment of Interoceptive Awareness | 16 weeks after start of TENS treatment
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is an 8-scale state-trait questionnaire with 32 items to measure multiple dimensions of interoception by self-report.
Return to work | 8 weeks after randomization
  Number of patients who return to work part time or full time.
Return to work | 16 weeks after start of TENS treatment
  Number of patients who return to work part time or full time.

CONTACTS AND LOCATIONS:
Overall Officials: Paulin Andéll, MD, Principal Investigator — Göteborgs Universitet/Västra Götalands Regionen
Locations (1):
- Pain Centre, Department of Anaesthesiology and Intensive Care Medicine Östra, Sahlgrenska University Hospital, Region Västra Götaland, Gothenburg, Sweden